CLINICAL TRIAL: NCT04873908
Title: Comparison of the Effect of Proprioceptive Training Therapy or Modified Constraint-Induced Movement Therapy on Upper Extremity Physical Functions in Chronic Stroke Patients - A Randomized Controlled Study
Brief Title: Effects of Modified Constraint-Induced on Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assit Prof. Nuray Alaca, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-24/05
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Stroke; Rehabilitation
Keywords: Modified constraint-induced therapy; Proprioceptive Training; conventional rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional rehabilitation (Other)
  Interventions: Other: conventional rehabilitation
- Modified constraint-induced therapy (Experimental)
  Interventions: Other: modified constraint-induced therapy
- Proprioceptive Training (Experimental)
  Interventions: Other: Proprioceptive Training

INTERVENTIONS:
Other: modified constraint-induced therapy — Patients received conventional rehabilitation and modified constraint-induced therapy schedule
  Arms: Modified constraint-induced therapy
Other: Proprioceptive Training — Patients received conventional rehabilitation and Proprioceptive Training schedule
  Arms: Proprioceptive Training
Other: conventional rehabilitation — Patients received conventional rehabilitation schedule
  Arms: conventional rehabilitation

SUMMARY:
In the present study, it was aimed to compare the proprioception training applied in addition to conventional treatment and Modified Constraint-Induced Movement Therapy treatment in patients with chronic strokes and to investigate the effects on proprioception, spasticity, functional motor skills and daily living activities in the upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* Post stroke hemiparetic patients of six months
* spasticity ≤ Grade -3 on modified Ashworth scale
* those patients capable of extension of at least 10º each at Metacarpophalangeal (MCP), Proximal Interphalangeal (PIP) and Distal Interphalangeal (DIP) joints and 20º at wrist joint
* a score of 24 or higher on the Modified Mini-Mental State Examination
* no excessive pain in the affected upper limb, as measured by a score of 4 or higher on a 10-point visual analog scale

Exclusion Criteria:

* Patients with history of previous stroke,
* angina,
* uncontrolled hypertension, on medication that could impair neuromuscular performance,
* wrist or finger pathologies, significant visual or hearing impairment,
* balance problems which may compromise safety during sound upper limb constraint,
* unwilling to participate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment test | Score change after 6 weeks of intervention compared to baseline
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based upper extremity function. The maximum available score is 66 and The minimum available score is zero.The higher total score means better motor function in the arm
Action Research arm test | Score change after 6 weeks of intervention compared to baseline
  The Action Research Arm Test (ARAT) is a 19 item observational measure used by physical therapists and other health care professionals to assess upper extremity performance. The maximum available score from the 19 items was 57. The higher total score means better motor function in the arm
Motor Activity Log | Score change after 6 weeks of intervention compared to baseline
  Daily use of the affected upper extremity was assessed using Motor Activity Log. It is a self-statement questionnaire to determine the frequency and quality of movement in the upper extremity. Score range is 0-5, The higher total score means better motor function in the arm

SECONDARY OUTCOMES:
Modified Ashworth Scale | Score change after 6 weeks of intervention compared to baseline
  Modified Ashworth Scale was measure muscle spasticity. It is among the most commonly used scales for clinical and research purposes. The resistance against passive movement is evaluated on a scale of 0-4 points.The lower total score means better spasticity in the arm
thumb localizing test | Score change after 6 weeks of intervention compared to baseline
  A proprioception examination, called the 'thumb localizing test' (TLT), is described as a technique for testing 'limb localization'. With the patient's eyes closed, the examiner positions one of the patient's upper limbs (fixed limb) and asks him to pinch the thumb of that limb with the opposite thumb and index finger (reaching limb).It is evaluated on a 0-3 point scale. The lower the total score, the better the proprioceptive in the arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided